CLINICAL TRIAL: NCT03497572
Title: Seroprevalence, Multi-center, Phase IV Cross-sectional Study to Evaluate the Persistence of Anti-leptospira Antibody in Subjects Vaccinated With Spirolept® Vaccine
Brief Title: Seroprevalence Study to Evaluate the Persistence of Anti-leptospira Antibody in Subjects Vaccinated With Spirolept® Vaccine
Acronym: SPT-001
Status: Completed | Type: Observational
Sponsor: Imaxio (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-A01797-46
Record Dates: First submitted 2017-08-10; First posted 2018-04-13 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Leptospirosis
Keywords: Leptospirosis
MeSH Terms: conditions — Leptospirosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — IgG, GIT are studied on serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to assess antibody persistence induced by Spirolept® vaccination in subjects who received at least 4 doses (2 doses two weeks apart and 2 booster doses) and no more than a total of 8 doses (2 doses two weeks apart and 6 booster doses).

DETAILED DESCRIPTION:
This is a seroprevalence, phase IV, multi -center study to evaluate anti-Leptospira antibody persistence in subjects who have received at least the 2nd booster (4 vaccine doses) and no more than the 6th booster (8 vaccine doses) of Spirolept® vaccine.

The study will be conducted at the Occupational Health Centre of companies employing workers at risk of leptospirosis for their occupational activities. Study participants will be selected from the company Occupational Health Centre database where each employee is registered. All workers are regularly followed-up and their medical and vaccination history recorded. Subjects selection will occur according the number of booster doses received (having received at least the 2nd booster and no more than the 6th booster). After they have signed the informed consent form, subjects will be recruited into the study and if all inclusion and exclusion criteria are met they will be taken a blood sample.

Anti-leptospira IgG antibody will be measured by a validated ELISA. Other assay may be performed to further characterize anti-leptospira antibodies. Data on subject demographics, relevant medical history, vaccination dates, and blood collection will be recorded in an appropriate Case Report Form.

The study does not include any vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both genders aged 18 to 65 years
* High risk occupational subjects to leptospirosis having received at least 4 (2 initial doses and 2 booster doses) and no more than 8 (2 first doses and 6 booster doses) doses of Spirolept®
* Previous Spirolept® vaccination dates documented
* To be affiliated to a health insurance plan
* Having signed the informed consent form

Exclusion Criteria:

* Had an acute infection during the 3 weeks before study enrollment
* Subject with documented HIV or hepatitis A, B, C
* Immunosuppressive treatment (chemotherapy, corticosteroids > 20mg/day, biological agents)
* Subject with progressive malignancy requiring specific treatment
* Previous documented Leptospirosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at the Occupational Health Centre of companies employing workers at risk of leptospirosis for their occupational activities. Study participants will be selected from the company Occupational Health Centre database where each employee is registered. All workers are regularly followed-up and their medical and vaccination history recorded. Subjects selection will occur according the number of booster doses received (having received at least the 2nd booster and no more than the 6th booster).
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
ELISA immunoglobulin G (IgG) anti-leptospire | through study completion, an average of 8 months
  Proportion of subjects seropositive to ELISA IgG anti-leptospira (with cut-off antibody titer ≥ 20) at different time points after the last booster dose

SECONDARY OUTCOMES:
ELISA IgG geometric mean titer (GMTs) | through study completion, an average of 8 months
  Proportion of subjects seropositive to ELISA IgG anti-leptospira (with cut-off antibody titer ≥ 20) and GMTs at different time points according to demographic factors and vaccination scheme

OTHER OUTCOMES:
exploratory growth inhibition test (GIT) Test | through study completion, an average of 8 months
  Proportion of subjects with positive GIT (positive GIT: serum that provides ≥ 50% leptospira growth inhibition in the test)

CONTACTS AND LOCATIONS:
Overall Officials: Maryse Beder, MD, Principal Investigator — SIAAP; Simonetta Viviani, MD, Study Director — Imaxio
Locations (2):
- France (2):
  - SIAAP, Maisons-Laffitte
  - Mairie de Paris, Paris